CLINICAL TRIAL: NCT04767750
Title: Role of LncRNA H19 in The Regulation of IGF-1R Expression: A Possible Association Between Type 2 Diabetes and Hepatocellular Carcinoma
Brief Title: Role of LncRNA H19 in The Regulation of IGF-1R Expression
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Other Study IDs: MS.20.10.26
Record Dates: First submitted 2020-12-21; First posted 2021-02-23 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2021-02

CONDITIONS: Hepatocellular Carcinoma; Type 2 Diabetes; Cancer
Keywords: LncRNA H19; IGF-1R
MeSH Terms: conditions — Carcinoma, Hepatocellular; Diabetes Mellitus, Type 2; Neoplasms; Insulin-Like Growth Factor I, Resistance To

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — 5ml of peripheral blood samples will be collected
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- HCC patients: Measure lncRNA H19 and IGF-1R mRNA gene expression levels in the collected blood samples.
  Interventions: Other: Blood sample collection
- T2DM patients: Measure lncRNA H19 and IGF-1R mRNA gene expression levels in the collected blood samples.
  Interventions: Other: Blood sample collection
- HCC & T2DM patients: Measure lncRNA H19 and IGF-1R mRNA gene expression levels in the collected blood samples.
  Interventions: Other: Blood sample collection
- Controls: Measure lncRNA H19 and IGF-1R mRNA gene expression levels in the collected blood samples.
  Interventions: Other: Blood sample collection

INTERVENTIONS:
Other: Blood sample collection — 5ml of peripheral blood samples will be collected into tubes containing EDTA from all subjects and the following procedures will be performed:
  * Peripheral blood mononuclear cells (PBMCs) will be isolated from blood samples.
  * Total RNA extraction from PBMCs by Trizol reagent and spin column.
  * Reverse transcription to cDNA.
  * The expression levels of lncRNA H19, IGF-1R mRNA and GAPDH gene (control gene) will be determined by Real-Time Quantitative PCR

SUMMARY:
Hepatocellular carcinoma (HCC) is a common cancer that poses a heavy economic burden on the healthcare system. In Egypt, it is the most common cause of mortality and morbidity-related cancer. Diabetes mellitus (DM) is a metabolic disorder characterized by hyperglycemia. Cancer and type II diabetes (T2DM), the world's two most prevalent diseases, share many overlapping risk factors and predisposing pathological conditions. The exact mechanisms linking those two diseases are yet to be fully understood.

In this study, the investigators aim to assess the relationship between Long Non-Coding RNA (lncRNA) H19 and Insulin-Like Growth Factor 1 Receptor (IGF-1R) mRNA gene expressions in the blood samples of HCC & T2DM patients to investigate the probability of the presence of a pathophysiological link between HCC and DM that may become a therapeutic target for both diseases. To the investigator's knowledge, there is currently no human research study investigating both H19 and IGF-1R in both DM and cancer.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is a common cancer that poses a heavy economic burden on the healthcare system. It represents the fourth and sixth most common cancer in Egypt and worldwide respectively. Globally, HCC is the fourth most common cause of death from cancer. It was estimated to be responsible for nearly 9.1% of the total deaths in 2012 (746,000 deaths). In Egypt, it is the most common cause of cancer-related mortality, and morbidity (32.35% of the total cancer deaths, mortality data were derived from the World Health Organization (WHO)). The leading risk factor in developing HCC in Egypt is hepatitis C virus (HCV).

Diabetes mellitus (DM) is a metabolic disorder characterized by hyperglycemia, which may be caused by insufficient insulin secretion, insulin resistance, or augmented glucagon production. Cancer and type II diabetes (T2DM), The world's two most prevalent diseases, share many overlapping risk factors and predisposing pathological conditions. Although the T2DM-cancer co-existence has been noted for many decades, the exact mechanisms linking these diseases are yet to be fully understood.

Insulin-Like Growth Factor-1 Receptor (IGF-1R) is a member of the insulin and IGF family. It coordinates a complex downstream signaling network through which it plays essential roles in the regulation of cell growth, proliferation, and survival as well as in glucose homeostasis. IGF-1R plays a crucial role in many tumor-related courses, such as tumor growth and metastasis in addition to drug resistance. The IGF-1R dysregulated signaling pathways in cancer and DM have been reported to be controlled at different levels by non-coding RNAs.

Non-coding RNAs (ncRNAs) are a large category of RNAs that usually do not participate in protein encoding but have a wide range of biological functions through regulation of protein expression and functions. The two most researched classes of ncRNAs are microRNAs (miRNAs) and the long non-coding RNAs (lncRNAs). H19 is a lncRNA that is found to be overexpressed in many solid tumors including HCC. The relationship between H19 and IGF-1R expression levels in addition to the dysregulation of H19 in DM are still inconsistent in literature, warranting further investigations. Ghazal et al. noted that H19 levels are directly proportional to IGF-1R expression levels in women with endometriosis (Ghazal et al., 2015). This is conflicting with Farzi-Molan et al. who remarked the reverse relation between IGF-1R & H19 during the differentiation of Bone Marrow Mesenchymal Stem Cells (BMSCs) to neural cells

ELIGIBILITY:
• HCC cases (group I):

Inclusion criteria:

- Patients aged 40 years or older with a confirmed diagnosis of HCC through triphasic CT and/or dynamic MRI (European Association for the Study of the Liver, 2012).

Exclusion criteria:

* Patients who underwent previous cancer-directed treatment (radiation and/or chemotherapy).
* Patients with any other systemic disease (Renal disease, other primary tumors).

  * T2DM cases (group II):

Inclusion criteria:

- Clinically diagnosed T2DM patients aged 40 years or older frequenting Mansoura Specialized Medical Hospital.

Exclusion criteria:

* Patients with previous or current malignancies.
* Patients with diabetic complications (Diabetic retinopathy, neuropathy, nephropathy).
* Patients with other systemic diseases.

  * HCC & T2DM cases (group III):

Inclusion criteria:

- Patients aged 40 years or older with a confirmed diagnosis of HCC through triphasic CT and/or dynamic MRI and who are clinically diagnosed to have T2DM.

Exclusion criteria:

* Patients who underwent previous cancer-directed treatment (radiation and/or chemotherapy).
* Patients with any other systemic disease.

  • Controls (group IV):
* Apparently healthy, age, and gender-matched subjects.
* No history of malignant disease, diabetes, or HCV.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This case-control study will be conducted in the Department of Medical Biochemistry and Molecular Biology, Faculty of Medicine, Mansoura University. Blood samples will be obtained from 24 HCC patients and 24 HCC & T2DM patients at the Gastroenterology Center, Mansoura University as well as from 26 T2DM patients at the Specialized Medical Hospital, Mansoura University in the period from December 2020 to December 2021.
  The study will include 101 patients divided into 4 groups:
  Group I: 24 HCC patients Group II: 26 T2DM patients Group III: 24 HCC & T2DM patients Group IV: 27 age and gender-matched healthy control volunteers. Written informed consent will be obtained from all individuals.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-04-04 (Actual)

PRIMARY OUTCOMES:
Measurement of the gene expression levels of LncRNA H19 & IGF-1R mRNA, normalized to the housekeeping gene GAPDH expression level, in HCC and T2DM in comparison with healthy controls using Real-Time Quantitative PCR (by the 2^-ΔΔCT method). | baseline
  To assess if there is a correlation between lncRNA H19 and IGF-1R mRNA gene expressions in the blood samples of HCC & T2DM patients to investigate the probability of the presence of a pathophysiological link between HCC and DM:
  * To measure the IGF-1R mRNA and lncRNA H19 expression levels in HCC & T2DM patients in comparison with healthy controls.
  * To investigate whether lncRNA H19 and IGF-1R mRNA expression levels affect one another.
  * To compare IGF-1R and lncRNA H19 expression levels in HCC associated with T2DM patients in contrast with sole affection with HCC or T2DM.

CONTACTS AND LOCATIONS:
Overall Officials: Noura MS Shehabeldin, M.B.B.Ch, Principal Investigator — Faculty of Medicine, Mansoura University.; Mohamed AA Zahran, M.D., Study Director — Faculty of Medicine, Mansoura University.; Heba K Mohamed, M.D., Study Chair — Faculty of Medicine, Mansoura University.; Nora M Hussein, M.D., Study Chair — Faculty of Medicine, Mansoura University.; Ahmed Shehta, M.D., Study Chair — Gastroenterology Center, Mansoura University; Helmy Ezzat, M.D., Study Chair — Gastroenterology Center, Mansoura University
Locations (2):
- Egypt (2):
  - Gastroenterology Center, Mansoura University, Al Mansurah, Dakahliya
  - Specialized Medical Hospital, Mansoura University, Al Mansurah, Dakahliya

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chen B, Li J, Chi D, Sahnoune I, Calin S, Girnita L, Calin GA. Non-Coding RNAs in IGF-1R Signaling Regulation: The Underlying Pathophysiological Link between Diabetes and Cancer. Cells. 2019 Dec 14;8(12):1638. doi: 10.3390/cells8121638. PMID 31847392
- [Background] Chitnis MM, Yuen JS, Protheroe AS, Pollak M, Macaulay VM. The type 1 insulin-like growth factor receptor pathway. Clin Cancer Res. 2008 Oct 15;14(20):6364-70. doi: 10.1158/1078-0432.CCR-07-4879. PMID 18927274
- [Background] Ding J, Li C, Tang J, Yi C, Liu JY, Qiu M. Higher Expression of Proteins in IGF/IR Axes in Colorectal Cancer is Associated with Type 2 Diabetes Mellitus. Pathol Oncol Res. 2016 Oct;22(4):773-9. doi: 10.1007/s12253-016-0065-6. Epub 2016 May 2. PMID 27138191
- [Background] Fabbri M, Girnita L, Varani G, Calin GA. Decrypting noncoding RNA interactions, structures, and functional networks. Genome Res. 2019 Sep;29(9):1377-1388. doi: 10.1101/gr.247239.118. Epub 2019 Aug 21. PMID 31434680
- [Background] Farzi-Molan A, Babashah S, Bakhshinejad B, Atashi A, Fakhr Taha M. Down-regulation of the non-coding RNA H19 and its derived miR-675 is concomitant with up-regulation of insulin-like growth factor receptor type 1 during neural-like differentiation of human bone marrow mesenchymal stem cells. Cell Biol Int. 2018 Aug;42(8):940-948. doi: 10.1002/cbin.10960. Epub 2018 Mar 30. PMID 29512257
- [Background] Ferlay J, Soerjomataram I, Dikshit R, Eser S, Mathers C, Rebelo M, Parkin DM, Forman D, Bray F. Cancer incidence and mortality worldwide: sources, methods and major patterns in GLOBOCAN 2012. Int J Cancer. 2015 Mar 1;136(5):E359-86. doi: 10.1002/ijc.29210. Epub 2014 Oct 9. PMID 25220842
- [Background] Forner A, Reig M, Bruix J. Hepatocellular carcinoma. Lancet. 2018 Mar 31;391(10127):1301-1314. doi: 10.1016/S0140-6736(18)30010-2. Epub 2018 Jan 5. PMID 29307467
- [Background] Ghazal S, McKinnon B, Zhou J, Mueller M, Men Y, Yang L, Mueller M, Flannery C, Huang Y, Taylor HS. H19 lncRNA alters stromal cell growth via IGF signaling in the endometrium of women with endometriosis. EMBO Mol Med. 2015 Aug;7(8):996-1003. doi: 10.15252/emmm.201505245. PMID 26089099
- [Background] Global Burden of Disease Liver Cancer Collaboration; Akinyemiju T, Abera S, Ahmed M, Alam N, Alemayohu MA, Allen C, Al-Raddadi R, Alvis-Guzman N, Amoako Y, Artaman A, Ayele TA, Barac A, Bensenor I, Berhane A, Bhutta Z, Castillo-Rivas J, Chitheer A, Choi JY, Cowie B, Dandona L, Dandona R, Dey S, Dicker D, Phuc H, Ekwueme DU, Zaki MS, Fischer F, Furst T, Hancock J, Hay SI, Hotez P, Jee SH, Kasaeian A, Khader Y, Khang YH, Kumar A, Kutz M, Larson H, Lopez A, Lunevicius R, Malekzadeh R, McAlinden C, Meier T, Mendoza W, Mokdad A, Moradi-Lakeh M, Nagel G, Nguyen Q, Nguyen G, Ogbo F, Patton G, Pereira DM, Pourmalek F, Qorbani M, Radfar A, Roshandel G, Salomon JA, Sanabria J, Sartorius B, Satpathy M, Sawhney M, Sepanlou S, Shackelford K, Shore H, Sun J, Mengistu DT, Topor-Madry R, Tran B, Ukwaja KN, Vlassov V, Vollset SE, Vos T, Wakayo T, Weiderpass E, Werdecker A, Yonemoto N, Younis M, Yu C, Zaidi Z, Zhu L, Murray CJL, Naghavi M, Fitzmaurice C. The Burden of Primary Liver Cancer and Underlying Etiologies From 1990 to 2015 at the Global, Regional, and National Level: Results From the Global Burden of Disease Study 2015. JAMA Oncol. 2017 Dec 1;3(12):1683-1691. doi: 10.1001/jamaoncol.2017.3055. PMID 28983565
- [Background] Hashad D, Elbanna A, Ibrahim A, Khedr G. Evaluation of the Role of Circulating Long Non-Coding RNA H19 as a Promising Novel Biomarker in Plasma of Patients with Gastric Cancer. J Clin Lab Anal. 2016 Nov;30(6):1100-1105. doi: 10.1002/jcla.21987. Epub 2016 May 17. PMID 27184562
- [Background] Huang JY, Wang SY, Lin Y, Yi HC, Niu JJ. The Diagnostic Performance of lncRNAs from Blood Specimens in Patients with Hepatocellular Carcinoma: A Meta-Analysis. Lab Med. 2021 Jan 4;52(1):64-73. doi: 10.1093/labmed/lmaa050. PMID 32700735
- [Background] Ibrahim AS, Khaled HM, Mikhail NN, Baraka H, Kamel H. Cancer incidence in egypt: results of the national population-based cancer registry program. J Cancer Epidemiol. 2014;2014:437971. doi: 10.1155/2014/437971. Epub 2014 Sep 21. PMID 25328522
- [Background] European Association For The Study Of The Liver; European Organisation For Research And Treatment Of Cancer. EASL-EORTC clinical practice guidelines: management of hepatocellular carcinoma. J Hepatol. 2012 Apr;56(4):908-43. doi: 10.1016/j.jhep.2011.12.001. No abstract available. PMID 22424438
- [Background] Matouk IJ, DeGroot N, Mezan S, Ayesh S, Abu-lail R, Hochberg A, Galun E. The H19 non-coding RNA is essential for human tumor growth. PLoS One. 2007 Sep 5;2(9):e845. doi: 10.1371/journal.pone.0000845. PMID 17786216
- [Background] Pollak M. The insulin and insulin-like growth factor receptor family in neoplasia: an update. Nat Rev Cancer. 2012 Feb 16;12(3):159-69. doi: 10.1038/nrc3215. PMID 22337149
- [Background] Rashed WM, Kandeil MAM, Mahmoud MO, Ezzat S. Hepatocellular Carcinoma (HCC) in Egypt: A comprehensive overview. J Egypt Natl Canc Inst. 2020 Jan 16;32(1):5. doi: 10.1186/s43046-020-0016-x. PMID 32372179
- [Background] Raveh E, Matouk IJ, Gilon M, Hochberg A. The H19 Long non-coding RNA in cancer initiation, progression and metastasis - a proposed unifying theory. Mol Cancer. 2015 Nov 4;14:184. doi: 10.1186/s12943-015-0458-2. PMID 26536864
- [Background] Villanueva A. Hepatocellular Carcinoma. N Engl J Med. 2019 Apr 11;380(15):1450-1462. doi: 10.1056/NEJMra1713263. No abstract available. PMID 30970190
- [Background] Ye Y, Guo J, Xiao P, Ning J, Zhang R, Liu P, Yu W, Xu L, Zhao Y, Yu J. Macrophages-induced long noncoding RNA H19 up-regulation triggers and activates the miR-193b/MAPK1 axis and promotes cell aggressiveness in hepatocellular carcinoma. Cancer Lett. 2020 Jan 28;469:310-322. doi: 10.1016/j.canlet.2019.11.001. Epub 2019 Nov 6. PMID 31705929
- [Background] Zhang N, Geng T, Wang Z, Zhang R, Cao T, Camporez JP, Cai SY, Liu Y, Dandolo L, Shulman GI, Carmichael GG, Taylor HS, Huang Y. Elevated hepatic expression of H19 long noncoding RNA contributes to diabetic hyperglycemia. JCI Insight. 2018 May 17;3(10):e120304. doi: 10.1172/jci.insight.120304. eCollection 2018 May 17. PMID 29769440
- [Background] Zhao M, Wang H, Chen J, Xi Y, Wang F, Huo C, Li W, Chu Y, Xu P, Huang Q, Bu S. Expression of long non-coding RNA H19 in colorectal cancer patients with type 2 diabetes. Arch Physiol Biochem. 2021 Jun;127(3):228-234. doi: 10.1080/13813455.2019.1628068. Epub 2019 Jun 22. PMID 31232113
- See also: Abudeif, A. (2019) 'Epidemiology and Risk Factors of Hepatocellular Carcinoma in Egypt', Sohag Medical Journal. Sohag University; Faculty of Medicine, 23(3), pp. 8-12. — https://smj.journals.ekb.eg/article_56178.html